CLINICAL TRIAL: NCT07242131
Title: Comparison of the Efficacy of Oral Contraceptive, Progesterone, and Inositol Use in Regulating Menstrual Cycles in Patients With Polycystic Ovary Syndrome (PCOS)
Brief Title: Efficacy of Oral Contraceptive, Progesterone, and Inositol on Menstrual Regulation in PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ad-PCOS-2
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic Ovary Syndrome; Menstrual Cycle; Didrogesterone
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Contraceptives, Oral, Combined; Ethinyl Estradiol; drospirenone; Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral Contraceptive Group (Active Comparator): Participants in this group will receive a combined oral contraceptive containing ethinylestradiol 0.03 mg and drospirenone 3 mg once daily for 21 days per cycle, followed by a 7-day pill-free interval, for 6 months. This arm serves as the active comparator to evaluate the relative efficacy of progesterone and myo-inositol therapy in menstrual regulation among women with PCOS.
  Interventions: Drug: Combined Oral Contraceptive (Ethinylestradiol 0.03 mg + Drospirenone 3 mg)
- Inositol Group (Experimental): Participants will receive oral inositol 2g/day for 6 months. This arm will assess the ability of myo-inositol to restore ovulatory cycles, improve ovarian morphology, and reduce hyperandrogenic symptoms in PCOS compared with oral contraceptive and progesterone groups.
  Interventions: Dietary Supplement: Inositol mid-level volume
- Progesterone (Didrogesterone) Group (Experimental): Participants will receive oral didrogesterone 10 mg twice daily from day 15 to day 25 of each menstrual cycle for 6 months. The efficacy of didrogesterone in restoring regular menstrual cycles and improving ovarian morphology will be compared with the oral contraceptive and myo-inositol groups.
  Interventions: Drug: Dydrogesterone Pill

INTERVENTIONS:
Drug: Combined Oral Contraceptive (Ethinylestradiol 0.03 mg + Drospirenone 3 mg) — Participants will receive one tablet daily for 21 consecutive days, followed by a 7-day pill-free interval, for a total of 6 months. Used as the standard treatment arm for menstrual regulation in PCOS.
  Arms: Oral Contraceptive Group
Dietary Supplement: Inositol mid-level volume — Participants will receive oral inositol 2 g/day for 6 months to assess its effects on ovulatory function, menstrual cycle regulation, and reduction of hyperandrogenic symptoms.
  Arms: Inositol Group
Drug: Dydrogesterone Pill — Participants will receive oral didrogesterone 10 mg twice daily from day 15 to day 25 of each menstrual cycle for 6 months (cyclic regimen).
  This arm evaluates the efficacy of oral didrogesterone monotherapy in restoring regular menstruation, improving ovarian morphology, and alleviating hyperandrogenic symptoms in women with PCOS, compared with inositol and oral contraceptive.
  Arms: Progesterone (Didrogesterone) Group

SUMMARY:
This cross-sectional study aims to compare the effectiveness of oral contraceptives, oral progesterone (didrogesterone), and inositol in regulating menstrual cycles among women diagnosed with polycystic ovary syndrome (PCOS).

PCOS is a common endocrine disorder affecting reproductive-aged women and is associated with menstrual irregularities, hyperandrogenism, and polycystic ovarian morphology. While oral contraceptives are the mainstay of treatment, their use may be contraindicated in patients with cardiovascular risk factors, liver dysfunction, or in those who desire pregnancy.

This study investigates whether oral progesterone and myo-inositol can serve as effective and safer alternatives for menstrual regulation and improvement of ovarian morphology and hyperandrogenic symptoms.

A total of 150 women aged 15-40 years with a diagnosis of PCOS will be enrolled and divided into three equal groups:

Group 1: Oral contraceptive users

Group 2: Oral progesterone users

Group 3: Inositol users The study will assess changes in menstrual regularity, ovarian morphology (via ultrasound), and clinical features such as hirsutism and acne before and after treatment.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder affecting women of reproductive age and is characterized by chronic anovulation, hyperandrogenism, and polycystic ovarian morphology. It is one of the most prevalent causes of infertility and is frequently associated with metabolic abnormalities such as insulin resistance, obesity, and dyslipidemia.

The primary treatment goal in PCOS is to restore regular ovulatory cycles, improve ovarian morphology, and reduce hyperandrogenic symptoms such as hirsutism and acne.

Combined oral contraceptives (COCs) are the first-line pharmacological option for cycle regulation in PCOS; however, their use is contraindicated in women with risk factors such as smoking, thromboembolic disorders, severe hepatic dysfunction, uncontrolled hypertension, or a history of breast cancer. Additionally, COCs are not suitable for women who desire pregnancy in the near future.

Therefore, alternative treatments that can effectively regulate menstrual cycles without suppressing fertility or inducing metabolic risks are clinically relevant.

This study aims to compare the effects of oral contraceptives, oral progesterone, and myo-inositol on menstrual regulation and ovarian morphology in women diagnosed with PCOS.

A total of 150 women aged 15-40 years who meet the ESHRE/ASRM (Rotterdam) diagnostic criteria for PCOS will be enrolled at the Department of Obstetrics and Gynecology, İzmir Bakırçay University Çiğli Training and Research Hospital. Participants will be randomly assigned to one of three groups (n=50 per group):

Group 1: Oral contraceptive users

Group 2: Oral progesterone users (didrogesterone 10 mg, twice daily, cyclic regimen)

Group 3: Inositol users (2 g/day)

Clinical parameters including menstrual regularity, body mass index, hirsutism score, acne grade, and ovarian morphology (assessed via transvaginal or transabdominal ultrasonography) will be recorded at baseline and follow-up visits.

The primary outcome will be restoration of regular menstrual cycles. Secondary outcomes will include changes in ovarian morphology, reduction of hyperandrogenic symptoms, and treatment tolerability.

Data will be analyzed using appropriate parametric or non-parametric statistical tests, with significance set at p<0.05.

All patient data will be anonymized, and participation will be voluntary following written informed consent. The study has been approved by the İzmir Bakırçay University Non-Interventional Clinical Research Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 to 40 years.
* Diagnosed with polycystic ovary syndrome (PCOS) according to the ESHRE/ASRM (Rotterdam) criteria (presence of at least two of the following: oligo/anovulation, clinical or biochemical hyperandrogenism, polycystic ovarian morphology).
* No significant comorbid systemic disease.
* Willingness to participate and ability to provide written informed consent.
* Regular follow-up availability for at least 6 months.

Exclusion Criteria:

* Known hepatic, renal, cardiovascular, or endocrine disorders other than PCOS.
* Pregnancy or current use of hormonal therapy within the past 3 months.
* History of thromboembolic disease, breast cancer, or other contraindications to hormonal treatment.
* Inability to adhere to follow-up visits or treatment regimen.
* Severe cognitive or communication impairment that prevents proper consent or data collection.
* Known allergy or hypersensitivity to any component of the study drugs.
* Participation in another interventional study within the past 3 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Restoration of Regular Menstrual Cycles | Baseline and at 6 months
  Evaluation of the proportion of participants who achieve restoration of regular menstrual cycles (defined as cycle length between 25-35 days for at least three consecutive cycles) after 6 months of treatment.

SECONDARY OUTCOMES:
Change in Ovarian Morphology | Baseline and at 6 months
  Assessment of changes in ovarian morphology via transvaginal or transabdominal ultrasonography, including ovarian volume and follicle count, compared with baseline.
Change in Serum Hormone Levels | Baseline and at 6 months
  Comparison of baseline and post-treatment serum levels of luteinizing hormone (LH), follicle-stimulating hormone (FSH), total testosterone, and estradiol to evaluate endocrine response to each treatment.
Patient Treatment Satisfaction | After 6 months of treatment
  Self-reported patient satisfaction and tolerability using a 5-point Likert scale evaluating ease of use, perceived effectiveness, and side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University, Izmir, Menemen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the findings of this study will be made available to qualified researchers upon reasonable request. Data will include demographic information, treatment group, and primary/secondary outcome measures. Personally identifiable information will be removed to ensure participant confidentiality.
  Data will be available after publication of the main results and upon approval by the principal investigator and the İzmir Bakırçay University Ethics Committee. Requests for access should be directed to the corresponding author via institutional email.
Supporting Information: Study Protocol, CSR
Time Frame: From 6 months after publication to 5 years post-publication.
Access Criteria: Access will be granted to researchers with methodologically sound proposals for academic and non-commercial purposes, following signing of a data access agreement.